CLINICAL TRIAL: NCT03714802
Title: Modified T-Stenting With Szabo Technique Versus T-Stenting for Bifurcation Lesions in Coronary Heart Diseases: SZABO Trial
Brief Title: Modified T-Stenting With Szabo Technique Versus T-Stenting for Bifurcation Lesions in Coronary Heart Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Professor Ge, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZABO Trial
Record Dates: First submitted 2018-09-21; First posted 2018-10-22 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2018-10

CONDITIONS: Coronary Artery Disease
Keywords: bifurcation lesion; percutaneous coronary intervention; Szabo; T-stenting
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Szabo T-Stenting Technique (Experimental): Patients received 2-stents implantation guided with Szabo technique in bifurcation lesion.
  Interventions: Procedure: Szabo T-Stenting Technique; Procedure: T-Stenting Technique
- T-Stenting Technique (Placebo Comparator): Patients received 2-stents implantation guided with T-stenting technique in bifurcation lesion.
  Interventions: Procedure: Szabo T-Stenting Technique; Procedure: T-Stenting Technique

INTERVENTIONS:
Procedure: Szabo T-Stenting Technique — 2-stent strategy was performed using modified T-stenting with Szabo technique in bifurcation lesions. First, stent was implanted in the side branch with Szabo technique. Then, stent was implanted in the main branch. Finally, kissing balloon inflation was performed.
Procedure: T-Stenting Technique — 2-stent strategy was performed using traditional T-stenting technique in bifurcation lesions. First, stent was implanted in the side branch with angiographic guidance. Then, stent was implanted in the main branch. Finally, kissing balloon inflation was performed.

SUMMARY:
The study will compare clinical outcomes of modified T-stenting with Szabo technique with T-stenting for bifurcation lesions in coronary heart diseases.

DETAILED DESCRIPTION:
Accurate deployment of stents in ostial lesions is difficult with traditional angiographic guidance. Szabo technique, which used a second angioplasty guide wire to anchor the stent by passing the proximal end of the anchor wire through the last cell of the stent, demonstrated accurate placement of the stents in ostial locations. In bifurcation lesions, 2-stent strategy positioning with Szabo technique was not investigated. Modified T-stenting with Szabo technique may improve prognosis of bifurcation lesions through reducing stents overlap. There is no clinical trial focuses on the effect and outcome of Szabo technique for coronary artery bifurcation lesions in contrast with conventional strategy.

In this study, the authors choose the closest 2-stent strategy, T-stenting, as control. We hope to determine whether a planned Szabo 2-stent technique is superior to T-stenting for patients with bifurcation lesions.

Patients with bifurcation lesions will be randomly assigned to receive Szabo 2-stent technique or T-stenting strategy. Clinical outcomes and imaging assessment will be used to estimate their effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least ≥18 years of age.
* Lesions are eligible for percutaneous coronary intervention (PCI).
* Patient has stable/unstable angina or myocardial infarction (MI).
* Bifurcation lesions (Medina 1,1,1/0,1,1/1,0,1) without left main ostial lesions.
* Downstream lesions could be covered by two stents.
* Diameter of vessel ≥2.25mm
* Diameter stenosis in main vessel and side branch ≥ 50% by visual estimation.

Exclusion Criteria:

* Severe tortuosity or calcification affected procedural success.
* Patient was allergic to the study stent or protocol-required concomitant medications.
* Patient is intolerable to dual anti-platelet therapy.
* Patient has any other serious medical illness that may reduce life expectancy to<12 months.
* Patient is a woman who is pregnant or nursing.
* Patient has a planned procedure that may cause non-compliance with the protocol or confound data interpretation.
* Patient is participating in another clinical trial that has not reached its primary endpoint within 24 months after the index procedure.
* Coronary restenosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiac death, nonfatal myocardial infarction and target lesion revascularization | 1 year after coronary angiography
  record in follow-up

SECONDARY OUTCOMES:
rate of all cause death | 30 days and 12 months after primary angiography
  Recorded in follow-up
rate of cardiac death rate | 30 days and 12 months after primary angiography
  Recorded in follow-up
rate of recurrent myocardial infarction rate | 30 days and 12 months after primary angiography
  Recorded in follow-up
rate of target vessel revascularization rate | 30 days and 12 months after primary angiography
  Recorded in follow-up
rate of stent thrombosis | 30 days and 12 months after primary angiography
  Recorded in follow-up
residual stenosis degree | Immediately after stent implantation and 12 months after primary angiography
  Measured through intravenous ultrasound
residual stenosis of side branch | Immediately after stent implantation and 12 months after primary angiography
  Measured through angiography
late lumen loss | index procedure and 12 months follow up
  Measured through intravenous ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Professor, Principal Investigator — Shanghai Zhongshan Hospital Fudan University
Locations (2):
- China (2):
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided